CLINICAL TRIAL: NCT03288064
Title: Effects of Corinthian Currant Supplementation on Redox Status, Inflammatory Markers, and Performance During Prolonged Exercise
Brief Title: Ergogenic and Antioxidant Effects of Corinthian Currant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Athanasios Z. Jamurtas, Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UTH2017AJCD
Record Dates: First submitted 2017-09-17; First posted 2017-09-19 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Athletic Performance; Oxidative Stress; Inflammation
Keywords: raisins; carbohydrates; antioxidant capacity; substrate oxidation; prolonged cycling
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Corinthian currant supplementation (Experimental): Corinthian currant supplementation: 1.5 g CHO/kg BW prior to exercise
  Interventions: Dietary Supplement: Corinthian currant
- Glucose supplementation (Experimental): Glucose drink (Top Star 100, Esteriplas, Portugal) supplementation: 1.5 g CHO/kg BW prior to exercise
  Interventions: Dietary Supplement: Glucose drink
- Water ingestion (Placebo Comparator): Water ingestion: 7 ml/kg BW prior to exercise
  Interventions: Dietary Supplement: Water ingestion

INTERVENTIONS:
Dietary Supplement: Corinthian currant — Supplementation of 1.5 g CHO/kg BW in the form of Corinthian currant prior to exercise
  Arms: Corinthian currant supplementation
Dietary Supplement: Glucose drink — Supplementation of 1.5 g CHO/kg BW in the form of glucose drink prior to exercise
  Arms: Glucose supplementation
Dietary Supplement: Water ingestion — Supplementation of 7ml/kg BW prior to exercise
  Arms: Water ingestion

SUMMARY:
The purpose of the present study is to investigate the effect of pre-exercise supplementation of Corinthian currant on metabolism, performance and blood redox status during, and after an acute bout of prolonged exercise.

Methods: Eleven healthy male adults (18 - 45y) performed an acute bout of prolonged cycling in a crossover fashion. Each bout consisted of a 90 min constant-intensity (70 - 75% VO2max) submaximal glycogen depletion trial, followed by a time trial (TT) to exhaustion (95% VO2max), with a wash out period of 2 weeks between bouts. During each experimental condition and 30 min prior to exercise, participants consumed an isocaloric (1.5 g CHO/kg body mass) amount of randomly assigned Corinthian currants, glucose drink, or water. Blood was drawn at baseline, 30 min after the supplement consumption (pre-exercise) and at 30, 60, 90 min of submaximal trial, after TT, and 1 h after the end of exercise (post TT), for the assessment of metabolic changes and redox status alterations.

DETAILED DESCRIPTION:
Aerobic exercise performance in events lasting more than one hour has been shown to improve with pre- or/and during-exercise consumption of carbohydrates (CHO) and athletes or recreationally exercised individuals are often advised to consume CHO before, and/or during exercise. The improvement in performance with CHO supplementation is due to the maintenance of blood glucose levels and the increased CHO availability for oxidation late in exercise that may preserve muscle glycogen. Apparently based on the above mechanisms, the dietary industry provides a wide variety of CHO supplements in different forms (sport drinks, sport gels, CHO bars, sport jellybeans, sport chews). Athletes at all levels use these supplements to optimize their performance during training or competitive events. However, these products are processed, and often expensive, in contrast with other natural foods that may provide an alternative for those preferring a healthier, though, equally effective choice.

Aerobic exercise and training relates with the production of reactive oxygen and nitrogen species (RONS), as indicated by the changes in the concentration of several by-products deriving from the oxidation of biomolecules, and the upregulation of antioxidant enzymes. Although RONS in low to moderate quantities are essential for optimized exercise performance and exercise-induced adaptations, yet, excessive production of RONS especially during exhaustive exercise, promote contractile dysfunction, muscle weakness and fatigue, and impaired recovery from exercise.Therefore, research has focused on nutritional strategies aimed at reducing these effects. There is evidence that treating with antioxidants, protects in part against free radicals-mediated damage in exercise. In regards with this prospective, the supplementation of antioxidants is a very common strategy to minimize RONS production and avoid the detrimental effects of oxidative stress in exercise. In the same way with CHO, natural foods could also provide an alternative antioxidant source for those seeking a more healthy option.

Corinthian currants or Corinthian raisins are small, dark purple colored, sun-dried vine products, produced from a special type of black grape (Vitis Vinifera L., var. Apyrena) and cultivated almost exclusively in the Southern of Greece. Corinthian currants are well known for their potential health benefits. They consist a high source of complex CHO (32.5% glucose, 32.1% fructose, 0.40% sucrose, 0.72% maltose), minerals (magnesium, iron, potassium, phosphorus, zinc) and vitamins (ascorbic acid, pyridoxine, riboﬂavin and thiamin) necessary for vitality, while they contain virtually no fat or cholesterol. Additionally, currants are considered as dried fruits with low to moderate glycemic index despite their high carbohydrate content. Therefore, Corinthian currant could be used as an alternative CHO source during exercise and provide a natural and healthy choice, equally effective to other commercial supplements on favorably affecting metabolism and/or improving performance.

Except for their high CHO content, Corinthian currants are also rich in polyphenols which are free radicals scavenging compounds and provide them with antioxidant properties. The rich antioxidant content renders Corinthian currant a potentially capable nutrient to boost an individual's antioxidant status in response to prolonged aerobic exercise. However, no study so far has addressed this potential role of Corinthian currants.

Therefore, the purpose of the present study was to investigate the effect of pre-exercise supplementation of Corinthian currants on metabolism and performance, as well as redox status in response to prolonged aerobic exercise. These responses were compared against glucose and water.

Eleven healthy well-trained male (n = 9) and female (n = 2) adults (18 - 45y) participated in the present cross over, randomized study. The participants visited the laboratory four times in total. During their ﬁrst visit, anthropometric characteristics assessment and baseline measurements were performed (body mass, standing height, percentage body fat, VO2max). Both the protocol for the assessment of VO2max, and the exercise protocol were performed on a cycle ergometer (Cycloergometer, Monark 834, ERGOMED C, Sweeden). During their second visit, the participants were randomly assigned to either Corinthian currant (1.5 g CHO/kg BW), or glucose drink (1.5 g CHO/kg BW), or water (6ml/kg BW) condition. After the assignment of the experimental condition, the participants performed the exercise protocol which consisted of 90 min of submaximal (70 - 75% VO2max) cycling, followed by a near maximal (95% VO2max) time trial to euxhastion. Fluid intake was kept constant at 7 ml/kg BW before the start of exercise, 3 ml/kg BW every 20 min during the 90-min exercise bout and 7 ml/kg BW within 15 min after the end of exercise. During their third and fourth visits, the participants repeated the experimental procedure after they had been assigned to one of the remaining two conditions. Between the first, second and third visit, there was a wash out period of two weeks. Blood samples were collected at baseline (before the CHO or water consumption), 30 min after CHO or water consumption (pre-exercise) and at 30 min, 60 min, 90 min of submaximal trial, after exhaustion (TT), and 1 h after the end of the exercise, for the assessment of GSH, catalase, uric acid , TAC, and TBARS.

ELIGIBILITY:
Inclusion Criteria:

* Normal BMI (18.5 - 24.99),absence of lower-limb musculoskeletal injury, absence of any metabolic disease, no drug/supplement consumption, and aerobic fitness (VO2max ≥ 40ml/kg/min at baseline testing).

Exclusion Criteria:

* Abnormal BMI (<18.5, ≥25), presence of lower-limb musculoskeletal injury, presence of any metabolic disease, no drug/supplement consumption, and aerobic fitness (VO2max < 40ml/kg/min at baseline testing).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2017-02-05 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Differences in time trial performance between conditions | After the 90 min submaximal exercise trial
  Participants performed an exercise protocol on a cycloergometer (Cycloergometer, Monark 834, ERGOMED C, Sweeden) consisted of 90 min of cycling at 70% - 75% VO2max, followed by a time trial (TT) at 95% VO2max to exhaustion or until the participants could not maintain a pace above 60 rpm. Gas exchange was monitored for the first 15 min until the desired steady state is established (70% - 75% VO2max), and every 25 min for 5 min thereafter.
Differences in glucose concentration (GLU) between conditions | At baseline, pre-exercise, 30 min, 60 min, 90 min of submaximal exercise trial, after exhaustion, 1 h post exercise
  Blood GLU concentration was assessed as a marker of human metabolism. Blood GLU concentration was estimated in a Clinical Chemistry Analyzer Z 1145 (Zafiropoulos Diagnostica, Athens, Greece) with commercially available kits (Zafiropoulos, Athens, Greece). Each sample is analyzed in duplicates.
Differences in lactate concentration (LA) between conditions | AAt baseline, pre-exercise, 30 min, 60 min, 90 min of submaximal exercise trial, after exhaustion, 1 h post exercise
  Blood LA concentration was assessed as a marker of human metabolism. Blood LA concentration was estimated in a Clinical Chemistry Analyzer Z 1145 (Zafiropoulos Diagnostica, Athens, Greece) with commercially available kits (Zafiropoulos, Athens, Greece). Each sample is analyzed in duplicates.
Differences in oxygen consumption (VO2) during exercise between conditions | During the first 15 min of submaximal exercise trial until the desired steady state of VO2 (70% - 75%) was established, and every 25 min for 5 min thereafter
  Cardiorespiratory changes were recorded throughout the entire exercise. Gas exchange was monitored using a gas analyzer (CareFusion, Viasis, Yorba Linda, USA).
Differences in carbon dioxide (CO2) during exercise between conditions | During the first 15 min of submaximal exercise trial until the desired steady state of VO2 (70% - 75%) was established, and every 25 min for 5 min thereafter
  Cardiorespiratory changes were recorded throughout the entire exercise. Gas exchange was monitored using a gas analyzer (CareFusion, Viasis, Yorba Linda, USA).
Differences in respiratory quotient (RQ) during exercise between conditions | During the first 15 min of submaximal exercise trial until the desired steady state of VO2 (70% - 75%) was established, and every 25 min for 5 min thereafter
  Cardiorespiratory changes were recorded throughout the entire exercise. Gas exchange was monitored using a gas analyzer (CareFusion, Viasis, Yorba Linda, USA).
Differences in ventilation (VE) during exercise between conditions | During the first 15 min of submaximal exercise trial until the desired steady state of VO2 (70% - 75%) was established, and every 25 min for 5 min thereafter
  Cardiorespiratory changes were recorded throughout the entire exercise. Gas exchange was monitored using a gas analyzer (CareFusion, Viasis, Yorba Linda, USA).
Differences in charbohydrates oxidation during exercise between conditions | During the first 15 min of submaximal exercise trial until the desired steady state of VO2 (70% - 75%) was established, and every 25 min for 5 min thereafter
  Cardiorespiratory changes were recorded throughout the entire exercise. Gas exchange was monitored using a gas analyzer (CareFusion, Viasis, Yorba Linda, USA).
Differences in fat oxidation changes during exercise between conditions | During the first 15 min of submaximal exercise trial until the desired steady state of VO2 (70% - 75%) was established, and every 25 min for 5 min thereafter
  Cardiorespiratory changes were recorded throughout the entire exercise. Gas exchange was monitored using a gas analyzer (CareFusion, Viasis, Yorba Linda, USA).
Differences in complete blood count (CBC) due to exercise between conditions | At baseline, pre-exercise, 30 min, 60 min, 90 min of submaximal exercise trial, after exhaustion, 1 h post exercise
  Assessment of CBC was performed in an automated hematological analyzer (Mythic 18, Orphee SA, Geneva, Switzerland).
Differences in reduced glutathione (GSH) (μmol/g Hb) due to exercise between conditions | At baseline, pre-exercise, 30 min, 60 min, 90 min of submaximal exercise trial, after exhaustion, 1 h post exercise
  GSH will be measured as a general index of oxidative stress. For GSH, 20 μL of erythrocyte lysate will be treated with 5% TCA mixed with 660 μL of 67 mM sodium potassium phosphate (pH 8.0) and 330 ΜL of 1 mM 5,5-dithiobis-2 nitrobenzoate. The samples will be incubated in the dark at room temperature for 45 min, and the absorbance will be read at 412 nm.
Differences in oxidized glutathione (GSSG) (μmol/g Hb) due to exercise between conditions | At baseline, pre-exercise, 30 min, 60 min, 90 min of submaximal exercise trial, after exhaustion, 1 h post exercise
  GSSG will be measured as a general index of oxidative stress. Blood collected will be treated with NEM. For the analysis, 50 μL of erythrocyte lysate will be treating with 5% TCA and neutralized up to pH 7.0-7.5. One microliter of 2-vinylpyridine will be added, and the samples will be incubated for 2 h. Sample will be treated with TCA and will be mixed with 600 μL of 143 mM sodium phosphate 100 ΜL of 3 mM NADPH, 100 ΜL of 10 mM 5,5-dithiobis-2-nitrobenzoate, and 194 μL of distilled water. After the addition of 1 μL of glutathione reductase, the change in absorbance at 412 nm will be read for 3 min.
Differences in thiobarbituric acid-reactive substances, TBARS (μM) due to exercise between conditions | At baseline, pre-exercise, 30 min, 60 min, 90 min of submaximal exercise trial, after exhaustion, 1 h post exercise
  TBARS will be measured as an index of lipid peroxidation. For TBARS determination, 100 μL of plasma will be mixed with 500 ΜL of 35% TCA and 500 μL of Tris-HCl (200 mM, pH 7.4) and will be incubated for 10 min at room temperature. One milliliter of 2 M Na2SO4 and 55 mM thiobarbituric acid solution will be added, and the samples will be incubated at 95O C for 45 min. The samples will be cooled on ice for 5 min and then will be vortexed after adding 1 mL of 70% TCA. The samples will be centrifuged at 15,000g for 3 min, and the absorbance of the supernatant will be read at 530 nm.
Differences in protein carbonyls, (PC) (nmol/mg pr) due to exercise between conditions | At baseline, pre-exercise, 30 min, 60 min, 90 min of submaximal exercise trial, after exhaustion, 1 h post exercise
  Changes in Protein carbonyls, PC (nmol/mg pr) Carbonyls will be measured as an index of protein oxidation. Protein carbonyls will be determined adding 50 μL of 20% TCA to 50 μL of plasma. Samples will be incubated in the dark at room temperature for 1 hour. The supernatant will be discarded, and 1 mL of 10% TCA will be added. The supernatant will be discarded, and 1 mL of ethanol-ethyl acetate will be added and centrifuged. The supernatant will be discarded, and 1 mL of 5 M urea will be added, vortexed, and incubated at 37C for 15 min. The samples will be centrifuged at 15,000g for 3 min at 4C, and the absorbance will be read at 375 nm.

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Z Jamurtas, Professor, Study Chair — University of Thessaly
Locations (1):
- School of Physical Education and Sport Science, University of Thessaly, Trikala, Thessaly, Greece

REFERENCES:
- [Result] Febbraio MA, Chiu A, Angus DJ, Arkinstall MJ, Hawley JA. Effects of carbohydrate ingestion before and during exercise on glucose kinetics and performance. J Appl Physiol (1985). 2000 Dec;89(6):2220-6. doi: 10.1152/jappl.2000.89.6.2220. PMID 11090571
- [Result] Jeukendrup AE, Killer SC. The myths surrounding pre-exercise carbohydrate feeding. Ann Nutr Metab. 2010;57 Suppl 2:18-25. doi: 10.1159/000322698. Epub 2011 Feb 22. PMID 21346333
- [Result] Chiou A, Panagopoulou EA, Gatzali F, De Marchi S, Karathanos VT. Anthocyanins content and antioxidant capacity of Corinthian currants (Vitis vinifera L., var. Apyrena). Food Chem. 2014 Mar 1;146:157-65. doi: 10.1016/j.foodchem.2013.09.062. Epub 2013 Sep 19. PMID 24176327
- [Result] Too BW, Cicai S, Hockett KR, Applegate E, Davis BA, Casazza GA. Natural versus commercial carbohydrate supplementation and endurance running performance. J Int Soc Sports Nutr. 2012 Jun 15;9(1):27. doi: 10.1186/1550-2783-9-27. PMID 22704463